CLINICAL TRIAL: NCT05426148
Title: A Study to Assess the Immunogenicity Consistency of Three Consecutive Batches of Commercial-scale of Recombinant Human Papillomavirus(HPV) Bivalent Vaccine (Escherichia Coli) in Healthy Female Subjects Aged 9-14 Years
Brief Title: Lot Consistency Clinical Trial of of Recombinant HPV Bivalent Vaccine in 9 to14 Years Old Healthy Female
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiamen Innovax Biotech Co., Ltd (Industry)
Collaborators: Jiangsu Province Centers for Disease Control and Prevention (Network); Dongtai City Centers for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HPV-PRO-010
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; Vaginal Intraepithelial Neoplasia; Vulvar Intraepithelial Neoplasia; Persistent Infection
Keywords: Human Papillomavirus Infection; Bivalent HPV Vaccine; Immunogenicity
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Persistent Infection; Papillomavirus Infections | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bivalent HPV Vaccine Consistency Lot 1 (Experimental): Biological/Vaccine: Participants would receive 2 doses of Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) intramuscularly at 0, 6 month.
  Interventions: Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) / Cecolin®
- Bivalent HPV Vaccine Consistency Lot 2 (Experimental): Biological/Vaccine: Participants would receive 2 doses of Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) intramuscularly at 0, 6 month.
  Interventions: Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) / Cecolin®
- Bivalent HPV Vaccine Consistency Lot 3 (Experimental): Biological/Vaccine: Participants would receive 2 doses of Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) intramuscularly at 0, 6 month.
  Interventions: Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) / Cecolin®

INTERVENTIONS:
Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) / Cecolin® — The bivalent HPV 16/18 vaccine was a mixture of two aluminum hydroxide adjuvant-absorbed recombinant L1 VLPs of HPV-16 and HPV-18 expressed in E. coli. A 0.5 ml dose of the bivalent HPV test vaccine comprised 40 μg of HPV-16 and 20 μg of HPV-18 L1 VLPs absorbed with aluminum adjuvant.
  Other Names: There is no other Intervention in this study

SUMMARY:
This study is to evaluate lot-lot consistency of Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) .

DETAILED DESCRIPTION:
This study is a mono-center, randomization, double-blind clinical trial in healthy Female subjects between 9 to 14. Under the premise of full informed consent, 540 subjects that meet the requirement of clinical trial in the age of 9-14 will be randomly divided into 3 groups in a ratio of 1:1:1 and injected 2 consecutive batches of Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) Cecolin® separately. The main outcome measures are the immunogenicity consistency and safety surveillance after inoculation according to prescribed immunization procedure.The total number of subjects should be ≥540 and ≤570.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged over 9 years old to 14 years old Female at the time of the first vaccine injection;
* 2. Statutory guardian of the subjects able to provide legal identification or the trustee able to provide the authorization certificate;
* 3. Judged as healthy and eligible for vaccination by the investigators through a selfreported medical history and some physical examinations;
* 4.Axillary temperature is below than 37.0 ℃;
* 5.Negative for urine pregnancy test.
* 6.The statutory guardian and trustee able to understand this study information and willing to comply with all study requirements(the statutory guardian or subject able to fill in the diary card and attend the follow-up on schedule).
* 7.Willing to participate in this study and sign informed consent form.

Exclusion Criteria:

Exclusion criteria for the first vaccination:

1. Administration of HPV Vaccine before the study;
2. Use of any investigational product or non-registered product (drug or vaccine)within 30 days preceding the first dose of the study vaccine or plan to use during the study period;
3. Received immunosuppressed, immunoregulation therapy or corticosteroid systemic therapy for more than 14 days in the 6 months before entry, except local treatment(such as ointment, eyedrops, inhalants or nasal sprays);
4. Administration of any immunoglobulin or blood products within 3 months preceding the first dose of the study vaccine,or plan to use during the study period;
5. Administration of any inactivated vaccines within 14 days preceding the first dose of the study or attenuated live vaccines within 21 days preceding the first dose of the study;
6. Had a fever (axillary temperature over 38°C) within 3 days or acute illness, or use systemic antibiotics or antiviral treatment within 5 days before vaccination;
7. Participate in any other clinical trial during the study period;
8. Immunodeficiency (such as HIV carriers), primary disease of important organs, malignant tumor, or any immune disease (such as systemic lupus erythematosus, rheumatoid arthritis, splenectomy or functional asplenia or other disease which might affect immune response), or other chronic diseases requiring treatment;
9. History of allergic disease or history of serious adverse events occurring after vaccination, such as allergy,urticaria, dyspnea, angioneurotic edema or abdominal pain;
10. Asthma that needed emergency treatment, hospitalization, oral or intravenous corticosteroid to keep stable in the past two years;
11. Combining another severe internal medicine disease(such as hypertension, cardiopathy,diabetes and hyperthyroidism);
12. Anormal coagulation function or coagulopathy diagnosed by doctor;
13. Epilepsy(not including febrile seizures under 2 years old, alcohol epilepsy within 3 years prior to abstinence and simple epilepsy that have not required treatment within 3 years prior to the study) ;
14. Anormal psychology or mind affecting the individual ability to obey the study requirements. Psychiatric disorders, not controlled in the past two years, required medication, or suicidal tendency in the past five years;
15. Other medical, psychological, social or occupational factors that, according to the investigators' judgment, might affect the individual ability to obey the protocol or sign the informed consent.

Exclusion criteria for second vaccination:

1. History of serious allergic reaction occurring after the first HPV vaccination;
2. History of serious adverse events following immunization caused by the first HPV vaccination;
3. Subject with new discovery or occurrence that does not meet the inclusion criteria, or conform to the exclusion criteria after the first HPV vaccination;
4. According to the judgment of the investigator, subject has newly discovered or emerging severe internal medicine disease, anormal coagulation function or coagulopathy that is not suitable for participating after the first HPV vaccination.

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Cecolin® is indicated for women to prevent the diseases caused by human papillomavirus (HPV) types 16 and/or 18, such as cervical cancer, cervical intraepithelial neoplasia Grade 2 or 3 (CIN2/3) and adenocarcinoma in-situ (AIS).
Enrollment: 540 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The Geometric Mean concentration (GMC) of anti-HPV16/18 IgG at at one month after the 2nd dose. | 7 months
  Measure anti-HPV16/18 IgG in serum samples at 7 month to evaluate the immunogenicity of the HPV vaccine.

SECONDARY OUTCOMES:
Seroconversion rate of anti-HPV16/18 IgG at one month after the 2nd dose. | 7 months
  Describe seroconversion rate of anti-HPV16/18 IgG one month after the last dose.
Measure solicited local adverse reactions within 7 days after each vaccination. | 7 days
Measure solicited systematic adverse reactions within 7 days after each vaccination. | 7 days
Measure unsolicited adverse reactions within 30 days after vaccination. | 30 days
Measure serious adverse events occurred throughout the study. | up to 7 months
Measure Potential Immune Mediated Diseases occurred throughout the study. | up to 7 months
  The Potential Immune Mediated Diseases refers to a disease of immune hyperfunction or immune deficiency caused by immune regulation disorder due to insufficient transmission of certain immune mediates, such as Guillain-Barre syndrome and thrombocytopenic purpura.

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (1):
- Dongtai City Center for Disease Control and Prevention Dongtai, Jiangsu, Dongtai, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No